CLINICAL TRIAL: NCT00422240
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group Study to Demonstrate the Efficacy and Safety of Adapalene/Benzoyl Peroxide Topical Gel Compared With Adapalene Topical Gel, 0.1%; Benzoyl Peroxide Topical Gel, 2.5% and Topical Gel Vehicle in Subjects With Acne Vulgaris
Brief Title: Study to Demonstrate the Efficacy and Safety of Adapalene/Benzoyl Peroxide Topical Gel in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.18087
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-10

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Adapalene; Benzoyl Peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Adapalene/Benzoyl Peroxide Gel (Experimental): Participants were treated with adapalene 0.1 % [weight by weight (W/W)]/benzoyl peroxide 2.5 % (W/W) gel topically daily in the evening for 12 Weeks.
  Interventions: Drug: Adapalene/Benzoyl Peroxide
- Adapalene Gel, 0.1% (Experimental): Participants were treated with 0.1% of adapalene gel topically daily in the evening for 12 Weeks.
  Interventions: Drug: Adapalene Gel, 0.1%
- Benzoyl Peroxide Gel 2.5% (Experimental): Participants were treated with 2.5% of benzoyl peroxide gel topically daily in the evening for 12 Weeks.
  Interventions: Drug: Benzoyl Peroxide Gel 2.5%
- Gel Vehicle (Placebo Comparator): Participants were treated with gel vehicle topically daily in the evening for 12 Weeks.
  Interventions: Drug: Gel Vehicle

INTERVENTIONS:
Drug: Adapalene/Benzoyl Peroxide — Adapalene 0.1 % [weight by weight (W/W)]/benzoyl peroxide 2.5 % (W/W) gel topically daily in the evening for 12 Weeks.
  Arms: Adapalene/Benzoyl Peroxide Gel
Drug: Adapalene Gel, 0.1% — 0.1% of adapalene gel topically daily in the evening for 12 Weeks.
  Arms: Adapalene Gel, 0.1%
Drug: Benzoyl Peroxide Gel 2.5% — 2.5% of benzoyl peroxide gel topically daily in the evening for 12 Weeks.
  Arms: Benzoyl Peroxide Gel 2.5%
Drug: Gel Vehicle — Participants were treated with gel vehicle topically daily in the evening for 12 Weeks.
  Arms: Gel Vehicle

SUMMARY:
This was a multi-center, randomized, double-blind, parallel group study with 12 weeks of treatment of acne vulgaris. Efficacy and safety evaluations were performed at Screening (safety only), Baseline and Weeks 1, 2, 4, 8 and 12. All Investigator's Global Assessment evaluators and lesion counters must be trained and approved by Galderma. The evaluator of a participant should remain the same during the study.

The primary objective was to demonstrate the superiority in efficacy and assess safety of adapalene/benzoyl peroxide topical gel (adapalene/benzoyl peroxide gel) versus adapalene topical gel, 0.1% (adapalene monad); benzoyl peroxide topical gel, 2.5% (benzoyl peroxide monad) and topical gel vehicle (gel vehicle) in the treatment of acne vulgaris for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of acne vulgaris with facial involvement.
* A minimum of 20 but not more than 50 inflammatory lesions
* A minimum of 30 but not more than 100 noninflammatory lesions
* A score of 3 (Moderate) on the Investigator's Global Assessment Scale

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1668 (Actual)
Dates: Start 2006-06-27 (Actual); Primary Completion 2007-07-12 (Actual); Study Completion 2007-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (1):
- Miller MD, San Antonio, Texas, United States

REFERENCES:
- [Background] Leyden JJ. A review of the use of combination therapies for the treatment of acne vulgaris. J Am Acad Dermatol. 2003 Sep;49(3 Suppl):S200-10. doi: 10.1067/s0190-9622(03)01154-x. PMID 12963896
- [Derived] Gold LS, Tan J, Cruz-Santana A, Papp K, Poulin Y, Schlessinger J, Gidner J, Liu Y, Graeber M; Adapalene-BPO Study Group. A North American study of adapalene-benzoyl peroxide combination gel in the treatment of acne. Cutis. 2009 Aug;84(2):110-6. PMID 19746769
- See also: Related Info — http://www.galderma.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1668 participants with acne vulgaris were randomized, administered and enrolled.
Period: Overall Study
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
Started | 415 | 420 | 415 | 418
Completed | 347 | 363 | 372 | 347
Not Completed | 68 | 57 | 43 | 71
Not completed — Lack of Efficacy | 1 | 2 | 0 | 1
Not completed — Adverse Event | 11 | 4 | 5 | 2
Not completed — Subject request | 21 | 17 | 18 | 30
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 31 | 32 | 19 | 34
Not completed — Other | 1 | 0 | 0 | 1
Not completed — Pregnancy | 3 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: ITT (Intent-to-Treat) Population included all treated participants.
Groups:
- Adapalene/Benzoyl Peroxide Gel: Participants were treated with adapalene 0.1 % (W/W)/benzoyl peroxide 2.5 % (W/W) gel topically daily in the evening for 12 Weeks.
- Total: Total of all reporting groups
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle | Total
Number analyzed (Participants) | 415 | 420 | 415 | 418 | 1668
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.7 (7.14) | 17.9 (5.40) | 18.4 (6.55) | 18.0 (6.09) | 18.2 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 217 | 207 | 222 | 856
  Male | 205 | 203 | 208 | 196 | 812
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 273 | 281 | 258 | 270 | 1082
  Black | 66 | 64 | 81 | 66 | 277
  Asian | 4 | 4 | 4 | 5 | 17
  Hispanic | 67 | 66 | 65 | 72 | 270
  Other | 5 | 5 | 7 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Success Rate 0 (Clear) or 1 (Almost Clear) on the Investigator Global Assessment (IGA) Scale at Week 12 (Last Observation Carried Forward)
Description: Success rate was defined as percentage of participants who achieved "Clear" or "Almost Clear" score on the IGA scale. IGA scale consisted of 5 grades (0-4) among which 0 = Clear (Minor, residual discoloration, no erythema or induration/papulation, no oozing/crusting), 1 = Almost clear (Trace, faint pink erythema with almost no induration/papulation and no oozing/crusting), 2 = Mild (Faint pink erythema with mild induration/papulation and no oozing/crusting), 3 = Moderate (Pink-red erythema with moderate induration/papulation and there may be some oozing/crusting.), 4 = Severe (Deep/bright red erythema with severe induration/papulation with oozing/crusting). All missing values were imputed by LOCF.
Time Frame: At Week 12
Population: ITT (Intent-To-Treat) Population included all treated participants. Here, Overall Number of Participants Analyzed = Participants with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- Adapalene/Benzoyl Peroxide Gel: Participants were treated with adapalene 0.1 % [weight by weight (W/W))]/benzoyl peroxide 2.5 % (W/W) gel topically daily in the evening for 12 Weeks.
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
Number analyzed (Participants) | 415 | 420 | 415 | 417
percentage of participants | 30.1 | 19.8 | 22.2 | 11.3

2. Primary Outcome: Change in Inflammatory Lesion Count From Baseline to Week 12
Description: Change in inflammatory lesion count from baseline to week 12 was reported. All missing values were imputed by LOCF.
Time Frame: Baseline to Week 12
Population: ITT Population included all treated participants.
Measure: Median (Inter-Quartile Range); unit: lesions
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
Number analyzed (Participants) | 415 | 420 | 415 | 418
lesions
  Baseline | 27.0 [23 to 35] | 27.0 [23 to 34] | 27.0 [23 to 34] | 27.0 [22 to 35]
  Change at Week 12 | -16.0 [-22 to -10] | -14.0 [-20 to -7] | -16.0 [-21 to -7] | -10.0 [-16 to -2]

3. Primary Outcome: Change in Noninflammatory Lesion Count From Baseline to Week 12
Description: Change in noninflammatory lesion count from baseline to week 12 was reported. All missing values were imputed by LOCF.
Time Frame: Baseline to Week 12
Population: ITT Population included all treated participants.
Measure: Median (Inter-Quartile Range); unit: lesions
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
Number analyzed (Participants) | 415 | 420 | 415 | 418
lesions
  Baseline | 44.0 [36 to 62] | 47.0 [37 to 61] | 46.0 [36 to 63] | 46.0 [36 to 62]
  Change at Week 12 | -24.0 [-35 to -13] | -22.0 [-34 to -11] | -20.0 [-32 to -7] | -14.0 [-25 to -1]

4. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts at Week 12
Description: The Inflammatory Lesion Count was the sum of papules and pustules. Percent change from Baseline was calculated as the values at Week 12 minus the value at Baseline divided by Baseline value * 100. All missing values were imputed by LOCF.
Time Frame: Baseline, Week 12
Population: ITT Population included all treated participants.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
Number analyzed (Participants) | 415 | 420 | 415 | 418
percent change | -55.33 (34.678) | -41.68 (41.855) | -47.61 (38.415) | -30.23 (41.661)

5. Secondary Outcome: Percent Change From Baseline in Noninflammatory Lesion Counts at Week 12
Description: The Noninflammatory Lesion Count was the sum of open comedones and closed comedones. Percent change from Baseline was calculated as the values at Week 12 minus the value at Baseline divided by Baseline value * 100. All missing values were imputed by LOCF.
Time Frame: Baseline, Week 12
Population: ITT Population included all treated participants.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
Number analyzed (Participants) | 415 | 420 | 415 | 418
percent change | -48.15 (35.428) | -40.75 (40.822) | -37.23 (39.758) | -23.22 (48.613)

6. Secondary Outcome: Percent Change From Baseline in Total Lesion Counts at Week 12
Description: The Total Lesion Count was the sum of Inflammatory, Noninflammatory Lesion Counts, Nodules and Cysts.
Time Frame: Baseline, Week 12
Population: ITT Population included all treated participants.
Measure: Mean (Standard Deviation); unit: percent change in lesions
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
Number analyzed (Participants) | 415 | 420 | 415 | 418
percent change in lesions | -49.97 (31.966) | -41.29 (36.133) | -41.23 (33.794) | -26.06 (38.714)

ADVERSE EVENTS:
Time Frame: From start of the study drug administration up to Week 12.
Description: Analysis was performed on safety population that included all participants who applied the study medication at least once.
Arm/Group | Adapalene/Benzoyl Peroxide Gel | Adapalene Gel, 0.1% | Benzoyl Peroxide Gel 2.5% | Gel Vehicle
All-Cause Mortality (participants affected / at risk) | 0/415 | 0/420 | 0/415 | 0/418
Serious Adverse Events (participants affected / at risk) | 2/415 | 3/420 | 0/415 | 1/418
Other Adverse Events (participants affected / at risk) | 44/415 | 51/420 | 29/415 | 34/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene/Benzoyl Peroxide Gel (N=415) | Adapalene Gel, 0.1% (N=420) | Benzoyl Peroxide Gel 2.5% (N=415) | Gel Vehicle (N=418)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene/Benzoyl Peroxide Gel (N=415) | Adapalene Gel, 0.1% (N=420) | Benzoyl Peroxide Gel 2.5% (N=415) | Gel Vehicle (N=418)
Dry skin (Skin and subcutaneous tissue disorders) | 28 (28) | 21 (21) | 9 (9) | 13 (13)
Nasopharyngitis (Infections and infestations) | 16 (16) | 30 (30) | 20 (20) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes